CLINICAL TRIAL: NCT04290299
Title: Endometrial Cancer Conservative Treatment (E.C.Co). A Multicentre Archive
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Cancer Institute, Naples (Other)
Responsible Party: Sponsor
Other Study IDs: 13/15 oss
Record Dates: First submitted 2020-02-27; First posted 2020-02-28 (Actual); Last update posted 2021-10-13 (Actual); Status verified 2021-10

CONDITIONS: Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Data collection — Cancer (response, relapse) and fertility (pregnancy, delivery) outcomes

SUMMARY:
Approximately one fourth of cases of endometrial cancer (EC) are diagnosed in premenopausal women, of whom approximately 40% wish to preserve their fertility. When arising in young women, EC usually presents with favorable prognostic features, as a focal, well differentiated endometrioid tumor, with minimal or absent myometrial invasion. This profile corresponds to the Type 1 EC, which correlates with the estrogen/progesterone receptor positive (ER+/PR+) pattern. On the other hand, these patients frequently present with clinical signs of a hyperestrogenism (chronic anovulation, infertility, obesity). Primary progestin therapy has been demonstrated to be effective in early well differentiated tumors and in poor operative candidates with response rates ranging from 58-100%.Currently, the therapeutic approach to an early stage EC consists of a staging laparotomy/laparoscopy, including a total abdominal hysterectomy and bilateral salpingo-oophorectomy (TAH-BSO), peritoneal washings, and lymphadenectomy (pelvic and aortic), depending on the pathological risk profile pre- and intraoperatively determined. Therefore, the current standard of surgical approach is preclusive of fertility.

The worldwide experience and data on conservative management of EC are, however, still limited. Most of reports based on cases retrospectively collected, harboring potential methodological bias, using different treatments and drugs, and with insufficient follow-up.

Some systematic reviews have been published in the last decade, trying to summarize the literature data. Therapeutic results seem to be promising with a regression rate of approximately 75% and relapse occurring in 25-40% of cases, with anecdotical reports of deaths of disease (DOD). The fertility outcome was, however, not satisfying with about 30% pregnancy rate in patients attempting to conceive, and an overall low rate of assisted reproductive techniques (ART) despite the subfertile clinical profile.Therefore, there is a need for a prospective, multicentre cooperative project able to systematically collect data from consecutive patients treated according to defined (not necessarily identical) protocols, concerning the oncological, as well as, the obstetrical outcomes. Moreover, this project could represent the "template" in which a pretreatment fertility counseling, psychological support, and definitive surgery are routinely included according to shared criteria.

DETAILED DESCRIPTION:
PURPOSE The goal of this research project is to learn more about the safety of conservatively treating EC and about subsequent fertility outcome.

PROJECT TYPE Observational (patient archive) - The project runs within the framework of Gynecologic Cancer InterGroup (GCIG), thus, participating Centres must belong to one of the qualified National groups.

PROJECT DESIGN Observational model: Cohort

TIME PERSPECTIVE Prospective

ENDPOINT CLASSIFICATION Cancer (response, relapse) and fertility (pregnancy, delivery) outcomes

INTERVENTIONS Data collection

OUTCOME MEASURES Primary outcome measures

* Proportion of complete regression
* Duration of response
* Frequency and pattern of relapse
* Frequency of metachronous ovarian cancer
* Tumor-related deaths

Secondary outcome measures

* Treatment related morbidity
* Frequency of spontaneous pregnancies
* Frequency of pregnancies after ART
* Pattern of residual disease on definitive surgical specimens

REQUIREMENTS FOR PATIENT REGISTRATION

* Informed consent to personal data processing
* Existence of an IRB-approved local protocol that allows conservative treatment to be performed or statement that such treatment is considered as a standard (please note that such protocols should be shared with the database owner National Cancer Institute of Naples).

TREATMENT Since this is a archive, treatment is not dictated by a protocol. However, treatment has to be administered according to a IRB-approved local protocol (except for the countries where conservative treatment can be given outside a IRB-approved study because considered as a standard procedure).

DURATION A first phase of three years is planned, eventually followed by further three years.

PUBLICATION POLICY Data generated are property of all investigators and will be object of publication after general agreement.

DATA TO BE COLLECTED

Patient enrollment and registration of data are made by appropriate eCRFs via the Clinical Trials Unit of National Cancer Institute of Naples (Study Data Center) website through the following steps:

1. go to http://www.usc-intnapoli.net;
2. select language;
3. click "Ask for authorization" to create your personal account;
4. fill and send the "authorization form";
5. make a screenshot of the "authorization form" and send it to l.sparavigna@istitutotumori.na.it;
6. enter into to the system using your credentials and click on "E.C.Co.";
7. click "the join request form";
8. wait for authorization (a verification message will be sent to your email address within 24-48 h);
9. enter into to the system using your credentials and click on "E.C.Co." for patient registration and/or updating.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent to personal data processing
* Existence of an IRB-approved local protocol that allows conservative treatment to be performed or statement that such treatment is considered as a standard (please note that such protocols should be shared with the database owner National Cancer Institute of Naples).

Exclusion Criteria:

-

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: Premenopausal women diagnosed with endometrial cancer (EC)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2015-09-15 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-04-08 (Estimated)

PRIMARY OUTCOMES:
Proportion of complete regression | 10 years
Duration of response | 10 years
Frequency of relapse | 10 years
Pattern of relapse | 10 years
Frequency of metachronous ovarian cancer | 10 years
Tumor-related deaths | 10 years

SECONDARY OUTCOMES:
Treatment related morbidity | 10 years
Frequency of spontaneous pregnancies | 10 years
Frequency of pregnancies after ART | 10 years
Frequency of residual disease on definitive surgical specimens | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Greggi, MD, Principal Investigator — National Cancer Institute of Naples
Locations (19):
- Cooperative Ovarian Cancer Group (COGI), Stanford, California, United States
- ANZGOG - Australia and New Zealand Gynecological Oncology Group, Sydney, Australia
- AGO-AUST Arbeitsgemeinschaft Gynaekologische Onkologie, Vienna, Austria
- EORTC - European Organization for Research and Treatment of Cancer, Brussels, Belgium
- Canada (2):
  - NCIC Clinical Trials Group (Canadian Cancer Society Research Institute), Ottawa
  - PMHC (Princess Margaret Hospital Consortium), Toronto
- SGOG (Shanghai Gynecologic Oncology Group), Shanghai, China
- NSGO (Nordic Society of Gynecologic Oncology), Copenhagen, Denmark
- GINECO - Group d'Investigateurs Nationaux pour l'Etude des Cancers Ovariens, Paris, France
- Germany (2):
  - AGO-De Arbeitsgemeinschaft Gynaekologische Onkologie Studiengruppe Ovarialkarzinom, Berlin
  - NOGGO (Nord-Ostdeutsche Gesellschaft für Gynäkologische Onkologie), Berlin
- ICORG - Ireland Cooperative Oncology Research Group, Dublin, Ireland
- MITO (Multicenter Italian Trials in Ovarian cancer and gynecologic malignancies), Naples, Italy
- Japan (2):
  - GOTIC - Gynecologic Oncology Trial and Investigation Consortium, Katō
  - JGOG - Japanese Gynecologic Oncology Group, Tokyo
- DGOG - Dutch Gynecologic Oncology Group, Amsterdam, Netherlands
- KGOG - Korean Gynecologic Oncology Group, Seoul, South Korea
- GEICO - Grupo Espanol de Investigacion en Cancer de Ovario, Madrid, Spain
- SGCTG (Scottish Gynaecological Cancer Trials Group), Edinburgh, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Data generated are property of all investigators and will be object of publication after general agreement.